CLINICAL TRIAL: NCT00391339
Title: Bryophyllum p. Versus Nifedipine for the Treatment of Premature Contractions
Brief Title: Bryophyllum vs. Nifedipine
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Weleda AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CI-C-64-Wel-06
Record Dates: First submitted 2006-10-19; First posted 2006-10-23 (Estimated); Last update posted 2006-10-23 (Estimated); Status verified 2006-10

CONDITIONS: Tocolysis
Keywords: Bryophyllum p.; Nifedipine; Tocolysis

INTERVENTIONS:
Drug: Bryophyllum p.

SUMMARY:
In a prospective, randomised study the efficacy and tolerability of bryophyllum p. (p.o) vs. nifedipine (p.o) will be proofed in a defined group of pregnant women with threatened preterm labour.

ELIGIBILITY:
Inclusion Criteria:

* Female

Exclusion Criteria:

* Bishop Score > 5

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140
Dates: Start 2006-11; Study Completion 2008-10

CONTACTS AND LOCATIONS:
Overall Officials: Roland Zimmermann, Prof. Dr. med., Principal Investigator — Department of Obstetrics, University Zuerich
Locations (1):
- Department of Obstetrics, University of Zuerich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Plangger N, Rist L, Zimmermann R, von Mandach U. Intravenous tocolysis with Bryophyllum pinnatum is better tolerated than beta-agonist application. Eur J Obstet Gynecol Reprod Biol. 2006 Feb 1;124(2):168-72. doi: 10.1016/j.ejogrb.2005.05.013. Epub 2005 Jul 26. PMID 16051414
- [Background] Gwehenberger B, Rist L, Huch R, von Mandach U. Effect of Bryophyllum pinnatum versus fenoterol on uterine contractility. Eur J Obstet Gynecol Reprod Biol. 2004 Apr 15;113(2):164-71. doi: 10.1016/S0301-2115(03)00370-1. PMID 15063954
- [Background] Vilaghy I. [Decreasing the rate of premature delivery with phytotherapy--results from general practice]. Ther Umsch. 2002 Dec;59(12):696-701. doi: 10.1024/0040-5930.59.12.696. German. PMID 12584959